CLINICAL TRIAL: NCT06272981
Title: Safety and Effectiveness Evaluation of the THERMOCOOL SMARTTOUCH™ SF Catheter With the TRUPULSE™ Generator for Treatment of Drug Refractory Symptomatic Paroxysmal Atrial Fibrillation (PAF)
Brief Title: A Study of the THERMOCOOL SMARTTOUCH Surround Flow (SF) Catheter With the TRUPULSE Generator for Treatment of Drug Refractory Symptomatic PAFOUS
Acronym: PulseSmart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI202308
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Pulsed Field (PF)/Radiofrequency (RF) Ablation System (Experimental): Participants with drug refractory symptomatic PAF who are candidates for atrial fibrillation ablation uses PF and RF energy to produce targeted intracardiac lesions for the treatment of atrial fibrillation.
  Interventions: Device: Pulsed Field (PF) /Radiofrequency (RF) Catheter ablation

INTERVENTIONS:
Device: Pulsed Field (PF) /Radiofrequency (RF) Catheter ablation — THERMOCOOL STSF catheter will be used in conjunction with TRUPULSE Generator to give PF ablation or RF ablation.

SUMMARY:
The purpose of this study is to demonstrate safety and effectiveness of the Biosense Webster (BWI) ablation system (THERMOCOOL SMARTTOUCH surround flow [STSF] catheter and TRUPULSE generator) when used for isolation of the atrial pulmonary veins (PVs) in treatment of participants with paroxysmal atrial fibrillation (PAF), an irregular heart rate that causing abnormal blood flow.

ELIGIBILITY:
Inclusion Criteria::

* Diagnosed with Symptomatic PAF (Physician's note indicating recurrent self-terminating AF). At least one (1) electrocardiographically documented AF episode within twelve (12) months prior to enrollment. Electrocardiographic documentation may include, but is not limited to, electrocardiogram (ECG), Holter monitor, or other electrocardiographical devices accepted by investigators
* Failed at least one (1) Class I or Class III Antiarrhythmic Drug (AAD) as evidenced by recurrent symptomatic AF or has intolerable side effects or is contraindicated to the Class I or Class III AAD
* Able and willing to comply with all pre-procedure, post-procedure, and follow-up testing and visit requirements
* Willing and capable of providing consent

Exclusion Criteria:

* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause (e.g., untreated documented obstructive sleep apnea and acute alcohol toxicity)
* Previous LA ablation or surgery
* Patients known to require ablation outside the PV region (atrioventricular reentrant tachycardia, atrioventricular nodal reentry tachycardia, atrial tachycardia, atrial flutter of unknown origin, ventricular tachycardia and Wolff-Parkinson-White)
* Previously diagnosed with persistent AF (> 7 days in duration)
* Severe dilatation of the LA (documented LAD >50mm antero-posterior diameter on imaging within 6 months prior to enrollment
* Documented left atrium (LA) thrombus within 48 hours prior to the index procedure by Transesophageal Echocardiography (TEE), or by Intracardiac Echocardiography (ICE) prior to transeptal puncture during procedure
* Documented severely compromised LVEF (LVEF <40%) by imaging within 6 months prior to enrollment
* Uncontrolled heart failure or New York Heart Association (NYHA) Class III or IV
* History of blood clotting, bleeding abnormalities or contraindication to anticoagulation (heparin, warfarin, or dabigatran)
* History of a documented thromboembolic event (including TIA) within the past 12 months, or history of a documented left atrial appendage (LAA) thrombus
* History of a documented symptomatic lacunar infarction within the past 12 months
* Previous PCI/MI within the past 2 months
* Coronary Artery Bypass Grafting (CABG) surgery within past 6 months
* Valvular surgery, cardiac surgery (e.g., ventriculotomy, atriotomy) or valvular cardiac (surgical or percutaneous) procedure
* Unstable angina pectoris within the past 6 months
* Anticipated cardiac transplantation, cardiac surgery or other major surgery within the next 12 months
* Significant pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
* Known significant PV anomaly that in the opinion of the investigator would preclude enrollment in this study
* Has known pulmonary vein stenosis
* Pre-existing hemi diaphragmatic paralysis
* Acute illness, active systemic infection or sepsis
* Presence of intracardiac thrombus, myxoma, tumor, interatrial baffle or patch or other abnormality that precludes catheter introduction or manipulation
* Severe mitral regurgitation (Regurgitant volume 60 mL/beat, Regurgitant fraction 50%, and/or Effective regurgitant orifice area 0.40cm^2)
* Presence of implanted pacemaker, Implantable Cardioverter-Defibrillator (ICD), recently implanted (within 6 months) LAAO device or other implanted metal cardiac device within the cardiac space that may interfere with the energy field created during the ablation procedure.
* Presence of a condition that precludes vascular access (such as IVC filter)
* Significant congenital anomaly or a medical problem that in the opinion of the investigator would preclude enrollment in this study
* Categorized as vulnerable population and requires special treatment with respect to safeguards of well-being
* Current enrollment in an investigational study evaluating another device or drug
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal), lactating, or who are of childbearing age and plan on becoming pregnant during the course of the clinical investigation
* Life expectancy less than 12 months
* History of massive hemorrhage within the past 6 months
* Presenting contra-indications for the devices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Primary Adverse Events (PAEs) | Within one week (7 days) post-procedure
  PAEs occurring within 7 days of an ablation which uses the BWI ablation system (including atrio-esophageal fistula and pulmonary vein stenosis occurring greater than 7 days of post ablation procedure) will be reported.
Rate of Freedom from Documented (Symptomatic and Asymptomatic) Atrial Arrhythmia (Atrial Fibrillation (AF), Atrial Tachycardia (AT) or Atrial Flutter (AFL) of Unknown Origin) within 91-365 Days Post Index Procedure | Within Day 91 to Day 365 post-procedure
  Rate of Freedom from documented (symptomatic and asymptomatic) atrial arrhythmia (AF, AT or AFL of unknown origin) within 91-365 days post index procedure will be reported. Freedom from atrial arrhythmia will be reported based on electrocardiographic data (greater than or equal to [>=30] seconds on arrhythmia monitoring device) during the effectiveness evaluation period (Day 91-Day 365) off antiarrhythmic therapy.

SECONDARY OUTCOMES:
Change from Baseline in Atrial Fibrillation Effect on Quality of Life (AFEQT) Total Score | Baseline, Month 12
  An overall AFEQT score ranges from 0 to 100. A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered). Therefore, a positive change in score corresponds to improvement in AF symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster, Inc. Clinical Trial, Study Director — Biosense Webster, Inc.
Locations (7):
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown
  - Canberra Heart Rhythm, Garran
  - Westmead Hospital, Westmead
- Canada (4):
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency